CLINICAL TRIAL: NCT01058863
Title: A Double-blind, Randomized, Placebo-controlled, 5-way Crossover, Multicenter, Single-dose, Dose-ranging Study to Compare the Efficacy and Safety of Albuterol Spiromax® and ProAir® HFA in Adult and Adolescent Subjects Ages 12 and Older With Persistent Asthma
Brief Title: A Dose-ranging Study to Evaluate Albuterol and Hydrofluoroalkane in Subjects Ages 12 and Older With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ABS-AS-201
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Albuterol Spiromax® 90 mcg (Experimental): A single dose of albuterol 90 mcg delivered with Spiromax®, an inhalation-driven, multi-dose dry powder inhaler. Placebo inhalers used to maintain the blind.
  Interventions: Drug: Albuterol Spiromax®; Other: Placebo Inhaler
- Albuterol Spiromax® 180 mcg (Experimental): A single dose of albuterol 180 mcg delivered with Spiromax®, an inhalation-driven, multi-dose dry powder inhaler (2 inhalations). Placebo inhalers used to maintain the blind.
  Interventions: Drug: Albuterol Spiromax®; Other: Placebo Inhaler
- ProAir® HFA 90 mcg (Active Comparator): A single dose of albuterol 90 mcg delivered with ProAir®, a 'press-and-breathe', metered-dose, aerosol inhaler. Placebo inhalers used to maintain the blind.
  Interventions: Drug: ProAir® HFA; Other: Placebo Inhaler
- ProAir® HFA 180 mcg (Active Comparator): A single dose of albuterol 180 mcg delivered with ProAir®, a 'press-and-breathe', metered-dose, aerosol inhaler (2 inhalations). Placebo inhalers used to maintain the blind.
  Interventions: Drug: ProAir® HFA; Other: Placebo Inhaler
- Placebo Inhaler (Placebo Comparator): Placebo delivered with Spiromax®, an inhalation-driven, multi-dose dry powder inhaler, and with ProAir®, a 'press-and-breathe', metered-dose, aerosol inhaler. Placebo inhalers used to maintain the blind.
  Interventions: Other: Placebo Inhaler

INTERVENTIONS:
Drug: Albuterol Spiromax® — Albuterol Spiromax® delivers 90 mcg albuterol per inhalation. Doses of 180 mcg require two inhalations. Intervention given as double-blind medication on 2 of 5 treatment days, once at 90 mcg and once at 180 mcg.
  Other Names: ProAir® RespiClick, Albuterol multi-dose dry powder inhaler (MDPI)
  Arms: Albuterol Spiromax® 180 mcg; Albuterol Spiromax® 90 mcg
Drug: ProAir® HFA — ProAir® HFA delivers 90 mcg of albuterol per inhalation. Doses of 180 mcg require two inhalations. Intervention given as double-blind medication on 2 of 5 treatment days, once at 90 mcg and once at 180 mcg.
  Other Names: albuterol HFA-MDI
  Arms: ProAir® HFA 180 mcg; ProAir® HFA 90 mcg
Other: Placebo Inhaler — Placebo delivered in both the Spiromax® and HFA inhalers to maintain the blind and also to support the placebo treatment arm.

SUMMARY:
This study is examining how well a dry powder inhaler (DPI) of albuterol medication works to help adult and adolescent subjects 12 years of age and older with persistent asthma to improve lung function.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent,
* Be between 12 years of age and older,
* Male or Female, females of non-child bearing potential or using reliable contraception
* Asthma for at least 6 months, FEV1 (forced expiratory volume in 1 second) between 50-80% of predicted value, and reversibility greater than or equal to 15% following 180 mcg albuterol
* Stable low dose of Inhaled Corticosteroids
* Non-smoker, 12 months smoking-free and <=10-pack years history
* Otherwise healthy
* Other criteria apply

Exclusion Criteria:

* Pregnant
* Allergic to albuterol or severe milk protein allergy
* Must not be on another trial for 30days.
* Other criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Study Leader, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (13):
- United States (13):
  - Teva Clinical Study Site, Huntington Beach, California
  - Teva Clinical Study Site, Rolling Hills Est., California
  - Teva Clinical Study Site, San Diego, California
  - Teva Clinical Study Site, Colorado Springs, Colorado
  - Teva Clinical Study Site, Margate, Florida
  - Teva Clinical Study Site, Miami, Florida
  - Teva Clinical Study Site, St Louis, Missouri
  - Teva Clinical Study Site, Skillman, New Jersey
  - Teva Clinical Study Site, Raleigh, North Carolina
  - Teva Clinical Study Site, Cincinnati, Ohio
  - Teva Clinical Study Site, Dayton, Ohio
  - Teva Clinical Study Site, Medford, Oregon
  - Teva Clinical Study Site, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 163 patients were screened and 72 patients were randomized. Most screening failures did not qualify for the study based on reversibility or spirometry criteria.
Groups:
- All Randomized Participants: Participants were randomized to one of ten treatment sequences, which indicated the order of the 5 single-dose treatments administered in this 5-way crossover study.
Period: Overall Study
Arm/Group | All Randomized Participants
Started | 72
Safety and ITT Populations | 71 (One patient was randomized in error and never received the study drug.)
Treated With Albuterol Spiromax® 90 mcg | 68
Treated With Albuterol Spiromax® 180 mcg | 68
Treated With ProAir® HFA 90 mcg | 70
Treated With ProAir® HFA 180 mcg | 68
Treated With Placebo Inhaler | 69
Completed | 68
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Sponsor requested withdrawal | 1
Not completed — Randomized in error | 1

BASELINE CHARACTERISTICS:
Population: Randomized and treated
Groups:
- Randomized Treated Participants: Participants were randomized to one of ten treatment sequences, which indicated the order of the 5 single-dose treatments administered in this 5-way crossover study.
Arm/Group | Randomized Treated Participants
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.78)
Age, Customized [Number; unit: participants]
  12 to <18 years | 3
  18 to 65 years | 64
  >65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54
  Black or African American | 16
  Asian | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Not Latino or Hispanic | 67
  Latino or Hispanic | 4
Height [Mean (Standard Deviation); unit: cm] | 169.1 (9.49)
Weight [Mean (Standard Deviation); unit: kg] | 89.6 (22.77)

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6)
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. The baseline for each study day was the average of the 2 pre-dose FEV1 measurements on that study day.
  The first baseline spirometry was obtained between 6-11 AM. The highest FEV1 value from two acceptable values was captured for calculation of the efficacy endpoints. Assessments were obtained at approximately 0.5 hours and immediately before dosing, and 5 minutes, 0.25, 0.50, 0.75, 1, 2, 3, 4, 5 and 6 hours after completion of dosing.
Time Frame: Day 1 up to Day 30
Population: Intent to treat population: randomized participants who received at least 1 dose of randomized study medication and had at least 1 post-baseline assessment
Measure: Mean (Standard Error); unit: L*hour
Arm/Group | Albuterol Spiromax® 90 mcg | Albuterol Spiromax® 180 mcg | ProAir® HFA 90 mcg | ProAir® HFA 180 mcg | Placebo Inhaler
Number analyzed (Participants) | 68 | 68 | 70 | 68 | 69
L*hour | 1.21 (0.224) | 1.39 (0.224) | 1.12 (0.223) | 1.33 (0.224) | 0.24 (0.224)
Statistical Analysis 1: Comparison: Albuterol Spiromax® 180 mcg vs Placebo Inhaler; Of interest was the mean difference between each active group and placebo at each dose level. Analyses were performed at the 2-sided 0.05 significance level in this sequence: Albuterol Spiromax 180 mcg versus placebo; Albuterol Spiromax 90 mcg versus placebo, ProAir HFA 180 mcg versus placebo, and ProAir HFA 90 mcg versus placebo. If a test was not significant, no further tests were done. This sequential procedure preserved the error rate for the family of tests at the 0.05 level; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; Fixed effects of baseline FEV1 as a covariate, sequence, treatment group, period, and center, and random effect for subject within sequence; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [0.88 to 1.42], Standard Error of Mean 0.136
Statistical Analysis 2: Comparison: Albuterol Spiromax® 90 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [0.70 to 1.24], Standard Error of Mean 0.136
Statistical Analysis 3: Comparison: ProAir® HFA 180 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.81 to 1.35], Standard Error of Mean 0.136
Statistical Analysis 4: Comparison: ProAir® HFA 90 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.61 to 1.15], Standard Error of Mean 0.136

2. Secondary Outcome: Baseline-adjusted Percent-Predicted Forced Expiratory Volume in 1 Second (PPFEV1) Area Under the Curve (AUC 0-6)
Description: Percent-predicted FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. Percent-predicted FEV1 is the expected FEV1 taking into account age, height, gender and race, as per the National Health and Nutrition Examination Survey III (NHANES III) reference values.
  The first baseline spirometry was obtained between 6-11 AM. The highest FEV1 value from two acceptable values was captured for calculation of the efficacy endpoints. Assessments were obtained at approximately 0.5 hours and immediately before dosing, and 5 minutes, 0.25, 0.50, 0.75, 1, 2, 3, 4, 5 and 6 hours after completion of dosing.
Time Frame: Day 1 up to Day 30
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % predicted * hour
Arm/Group | Albuterol Spiromax® 90 mcg | Albuterol Spiromax® 180 mcg | ProAir® HFA 90 mcg | ProAir® HFA 180 mcg | Placebo Inhaler
Number analyzed (Participants) | 68 | 68 | 70 | 68 | 69
% predicted * hour | 35.31 (4.497) | 41.05 (4.495) | 33.19 (4.461) | 40.68 (4.496) | 7.58 (4.482)
Statistical Analysis 1: Comparison: Albuterol Spiromax® 180 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; Fixed effects of baseline PPFEV1 as a covariate, sequence, treatment group, period, and center, and random effect for subject within sequence; Mean Difference (Final Values) = 33.47, 95% CI 2-sided [26.21 to 40.74], Standard Error of Mean 3.690
Statistical Analysis 2: Comparison: Albuterol Spiromax® 90 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — Significance at the 0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 27.73, 95% CI 2-sided [20.47 to 34.99], Standard Error of Mean 3.686
Statistical Analysis 3: Comparison: ProAir® HFA 180 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 33.10, 95% CI 2-sided [25.84 to 40.35], Standard Error of Mean 3.686
Statistical Analysis 4: Comparison: ProAir® HFA 90 mcg vs Placebo Inhaler; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance at the 0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 25.61, 95% CI 2-sided [18.36 to 32.85], Standard Error of Mean 3.680

3. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 up to Day 37
Population: Safety population of all randomized participants who received at least one dose of randomized study medication.
Measure: Number; unit: participants
Groups:
- All Randomized Participants: Participants were randomized to one of five treatment arms, which indicated the order of the 5 single-dose treatments administered in this 5-way crossover study.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 71
participants
  Any adverse event | 9
  Treatment-related AE | 0
  Withdrawn from study due to AEs | 0
  Any serious AEs | 0
  Treatment-related serious AE | 0
  Onset treatment for AE: Placebo Inhaler | 2
  Onset treatment for AE: Albuterol Spiromax 90mcg | 3
  Onset treatment for AE: Albuterol Spiromax 180mcg | 3
  Onset treatment for AE: ProAir HFA 90 mcg | 0
  Onset treatment for AE: ProAir HFA 180 mcg | 2

ADVERSE EVENTS:
Time Frame: Day 1 to Day 37
Arm/Group | Albuterol Spiromax® 90 mcg | Albuterol Spiromax® 180 mcg | ProAir® HFA 90 mcg | ProAir® HFA 180 mcg | Placebo Inhaler
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68 | 0/70 | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 3/68 | 3/68 | 0/70 | 2/68 | 2/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol Spiromax® 90 mcg (N=68) | Albuterol Spiromax® 180 mcg (N=68) | ProAir® HFA 90 mcg (N=70) | ProAir® HFA 180 mcg (N=68) | Placebo Inhaler (N=69)
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Localized infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.